CLINICAL TRIAL: NCT06895239
Title: Elbow Arthroplasty and Patient Reported Post-operative Activities
Acronym: EAA
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 900
Record Dates: First submitted 2024-08-09; First posted 2025-03-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Elbow Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who underwent Total elbow replacement from and after 2010 with a minimum of 6 months at a single institution will be studied retrospectively. The data required for the study will be collected prospectively. Patient demographic data will be collected through the Information team and electronic patient record. Surveys will include questions about whether they recalled the activities that were not recommended by the surgeons, oxford elbow scores and the type of activities they currently perform. Patients will be contacted by telephone after initial screening against inclusion and exclusion criteria, and subsequent questionnaires will be sent through post or by email, whichever the patient prefers. Patients who do not respond to the postal or email questionnaire will be contacted again by telephone.

DETAILED DESCRIPTION:
Total elbow arthroplasty is an increasingly common treatment for patients with destructive elbow pathology like osteoarthritis, rheumatoid arthritis, trauma and trauma sequelae. However, the revision rates and complication rates for elbow arthroplasty are relatively high when compared to hip and knee arthroplasty. Failure is commonly due to aseptic loosening that is a likely consequence of overloading of the implants. This has resulted in implant manufacturers and surgeons recommending long-term activity restrictions to patients post-operatively. There are no standardised post-operative guidelines after elbow arthroplasty as the evidence base in the literature is poor. More recent efforts have been made to rectify this global issue. Post-operative activity levels have been reviewed with regards to other joints like the knee, hip and shoulder. However, there is evidence that adherence to post-operative restrictions after hip arthroplasty can be expected in less than 75% of patients, and general patient non-compliance with instructions can be as high as 27.5% after all orthopaedic procedures. The investigators could only find one single publication regarding patient compliance with activity restrictions after elbow arthroplasty, and this was over a decade ago. An awareness of patient comprehension and compliance with post-operative activity restriction with help surgeons and allied health professionals counsel patients more effectively pre-operatively and post-operatively.

The purpose of our study is to determine the overall level of activity and percentage of patients participating in moderate demand and high demand activities. The authors would also explore patient recall of activity restrictions and correlate this with their current activity levels.

In the literature, data regarding the specific activities performed by patients after total elbow arthroplasty are lacking. Knowledge of patient understanding of postoperative restrictions, as well as their compliance, may help improve preoperative and postoperative counselling of patients undergoing total elbow arthroplasty and help us understand the true relationship between activity and mechanical failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had elbow arthroplasty (total or hemi) for any indication. Minimum 6 months follow-up.

Exclusion Criteria:

* Radial head replacement.
* Less than 6 months follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant who have had elbow replacement at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine what activities patients are undertaking after elbow arthroplasty | From the time of their surgery until now, a minimum of 6 months since surgery.
  Explore patient activity after elbow arthroplasty and their recollection of activity restrictions placed as part of the post-operative protocol as part of standard care.
Oxford Elbow Score | From the time of their surgery until now, a minimum of 6 months since surgery.
  Validated questionnaire. The Oxford Elbow Score has 12 items (questions) with 5 response options each. Each item response is scored 0 to 4, with 0 representing greater severity.
Elbow replacement surgery and activities performed after the operation | From the time of their surgery until now, a minimum of 6 months since surgery.
  Non-validated questionnaire regarding activities performed after operation to assist us to understand and convey to other patients about what activities people can do after elbow replacement, along with employment status, whether the participant has a physically demanding job and whether they are still taking medication for their replaced elbow joint.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarkadas PC, Throckmorton TQ, Dahm DL, Sperling J, Schleck CD, Cofield R. Patient reported activities after shoulder replacement: total and hemiarthroplasty. J Shoulder Elbow Surg. 2011 Mar;20(2):273-80. doi: 10.1016/j.jse.2010.06.007. Epub 2010 Oct 15. PMID 20951063
- [Result] Samdanis V, Manoharan G, Jordan RW, Watts AC, Jenkins P, Kulkarni R, Thomas M, Rangan A, Hay SM. Indications and outcome in total elbow arthroplasty: A systematic review. Shoulder Elbow. 2020 Oct;12(5):353-361. doi: 10.1177/1758573219873001. Epub 2019 Sep 12. PMID 33093874
- [Result] Kholinne E, Arya A, Jeon IH. Complications of modern design total elbow replacement. J Clin Orthop Trauma. 2021 May 15;19:42-49. doi: 10.1016/j.jcot.2021.05.008. eCollection 2021 Aug. PMID 34141570
- [Result] Macken AA, Prkic A, van Oost I, Spekenbrink-Spooren A, The B, Eygendaal D. Implant survival of total elbow arthroplasty: analysis of 514 cases from the Dutch Arthroplasty Registry. Bone Jt Open. 2023 Feb 21;4(2):110-119. doi: 10.1302/2633-1462.42.BJO-2022-0152.R1. PMID 37051858
- [Result] Badre A, King GJW. Primary total elbow arthroplasty. J Clin Orthop Trauma. 2021 Apr 20;18:66-73. doi: 10.1016/j.jcot.2021.04.015. eCollection 2021 Jul. PMID 33996451
- [Result] Dam WV, Meijering D, Stevens M, Boerboom AL, Eygendaal D. Postoperative management of total elbow arthroplasty: Results of a European survey among orthopedic surgeons. PLoS One. 2022 Nov 14;17(11):e0277662. doi: 10.1371/journal.pone.0277662. eCollection 2022. PMID 36374842
- [Result] Burden EG, Evans JP, Smith CD. Lifting limitations following elbow arthroplasty: A survey of British Elbow and Shoulder Society members. Shoulder Elbow. 2024 Oct;16(6):641-645. doi: 10.1177/17585732231170292. Epub 2023 Apr 20. PMID 39650263